CLINICAL TRIAL: NCT01783626
Title: Evaluation of Evodial Hemodialyzer Selectivity Modifications (Evodial +) - A Prospective, Monocenter, Open and Non-randomized Pilot Study
Brief Title: Evaluation of Evodial Hemodialyzer Selectivity Modifications (Evodial +)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Lundia AB (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1498
Record Dates: First submitted 2013-01-28; First posted 2013-02-05 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Evodial (Sham Comparator): Period I: HDF post dilution Total Volume 8 liters : 1 HD session (2nd HD of the week) Period II: HDF post dilution Total Volume 20 liters : 1 HD session (2nd HD of the week)
  Interventions: Device: Evodial
- Evodial+ Condition B1 (Experimental): Period I: HDF post dilution Total Volume 8 liters : 1 HD session (2nd HD of the week) Period II: HDF post dilution Total Volume 20 liters : 1 HD session (2nd HD of the week)
  Interventions: Device: Evodial+ Condition B1
- Evodial+ Condition B2 (Experimental): Period I: HDF post dilution Total Volume 8 liters : 1 HD session (2nd HD of the week) Period II: HDF post dilution Total Volume 20 liters : 1 HD session (2nd HD of the week)
  Interventions: Device: Evodial+ Condition B2
- Evodial+ Condition C (Experimental): Period I: HDF post dilution Total Volume 8 liters : 1 HD session (2nd HD of the week) Period II: HDF post dilution Total Volume 20 liters : 1 HD session (2nd HD of the week)
  Interventions: Device: Evodial+ Condition C

INTERVENTIONS:
Device: Evodial
  Arms: Evodial
Device: Evodial+ Condition B1
  Arms: Evodial+ Condition B1
Device: Evodial+ Condition B2
  Arms: Evodial+ Condition B2
Device: Evodial+ Condition C
  Arms: Evodial+ Condition C

SUMMARY:
Evodial +hemodialyzer consists of an evolution of the existing CE marked Evodial device, with respect to the hemodialyzer membrane removal characteristics. Different membrane prototypes configurations are proposed (3 versions in total), with the objective to modulate the hemodialyzer removal capacities (convective and adsorptive capacities).

Materials(including heparin grafted specifications) as well as the sterilization process are identical to the Evodial hemodialyzer. Based on available preclinical data , a clinical study is requested to document in vivo the different prototypes removal capacities with respect to middle Molecular Weight (MW) reference toxins such as b2 Microglobulin and collect data with regards to protein loss.

ELIGIBILITY:
Inclusion Criteria:

1. Anuric patient (diuresis<300ml) ,
2. ESRD patient treated for at least 3 months,
3. Patient treated in HDF post-dilution,
4. Vascular access functioning properly (Qb > 250 ml/min),
5. Patient aged 18 years or more,
6. Written consent to participate in the study (informed consent).

Exclusion Criteria:

1. Patient with pre-dialytic albuminemia <3.3 g/dl(Nephelometry assay)
2. Patient with known allergy to heparin or type II heparininduced thrombocytopenia (HIT type II);
3. Patient under guardianship;
4. Women pregnant or breast feeding;
5. Patient included in other studies that could interfere with the goals of the current study.
6. Patient that are not affiliated to the health system(beneficiary or dependent).
7. Patient with positive serology (HIV, Hepatitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Efficacy: Beta 2 Microglobulin elimination | Change from T0 (dialysis start) at T4 hours (dialysis stop)

SECONDARY OUTCOMES:
Efficacy: -Elimination of Myoglobin,alpha 1 Microglobulin, alpha amylase and Factor D | Change from T0 (dialysis start) at T 4hours (dialysis stop)
Efficacy:Profile of ultrafiltrated proteins | at T4 hours
Safety: Follow-up of all AEs/SAEs | during the study period
Safety: Measurement of Albumin loss | At T4 hours
Efficacy: Cumulative Purified volume (Kt) | At T4 hours
Safety: Total protein | Change from T0 and T4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Loughraieb, Study Director — Gambro Industries
Locations (1):
- Hôpital Louis-Pasteur (Cherbourg-Octeville), Cherbourg-Octeville, France